CLINICAL TRIAL: NCT01633944
Title: Phase 3, Double-Blind, Placebo-Controlled, Study to Evaluate the Analgesic Efficacy, Safety, and Tolerability of Buprenorphine HCl Buccal Film in Opioid-Naive Subjects With Chronic Lower Back Pain Requiring Opioid Analgesia
Brief Title: Efficacy Study to Evaluate Buprenorphine HCl Buccal Film in Opioid-Naive Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3409-308
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Low Back Pain
Keywords: CLBP; Chronic Low Back Pain; Chronic Pain; Back Pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Back Pain | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Twice Daily Dosing
  Interventions: Drug: Placebo
- Buprenorphine HCl Buccal Film (Experimental): Twice Daily Dosing
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine HCl Buccal Film at doses ranging from 75-600 mcg twice daily
  Other Names: BELBUCA; Buprenorphine HCl Buccal Film; BEMA Buprenorphine; EN3409
  Arms: Buprenorphine HCl Buccal Film
Drug: Placebo — Matching Placebo Buccal Film twice daily
  Other Names: Placebo Buccal Film; BEMA Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if buprenorphine hydrochloride (HCl) buccal film is effective in treating opioid-naive subjects, with moderate to severe chronic low back pain (CLBP), who require continuous around-the-clock (ATC) pain relief for an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe low back pain for ≥6 months
* Treating CLBP with a stable daily maintenance dose of non-opioid analgesic medication up to 10 mg morphine sulfate equivalents (MSE) per day for ≥4 weeks. (Additional as needed [PRN] non-opioid analgesic medications permitted on top of the stable daily maintenance dose of non-opioid analgesic)
* Stable health, as determined by Principal Investigator
* Are female who are practicing abstinence or using a medically acceptable form of contraception or have been post-menopausal, biologically sterile, or surgically sterile for more than 1 year
* Willing and able to comply with all protocol required visits and assessments

Exclusion Criteria:

* Current cancer related pain or received chemotherapy with 6 months of screening
* Receiving opioid analgesic medication >10 mg MSE per day within 28 days of screening
* Subjects with a history of other chronic painful conditions
* Reflex sympathetic dystrophy or causalgia, acute spinal cord compression, cauda equina compression, acute nerve root compression, meningitis, or discitis
* Allergy or contraindications to any opioid or acetaminophen
* Surgical procedure for relief of pain with 6 months
* Hypokalemia or clinically unstable cardiac disease, including: unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, or active myocardial ischemia
* QT interval corrected using Fridericia's formula (QTcF) of ≥450 milliseconds on the 12-lead electrocardiogram (ECG)
* History of long QT syndrome or a family member with this condition
* Moderate to severe hepatic impairment
* Moderate to severe renal impairment
* Current or past history of alcohol abuse
* Positive urine toxicology screen for drug of abuse
* History or abnormalities on physical exam, vital signs, electrocardiogram, or laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Todd Kirby, PhD, Study Director — Endo Pharmaceuticals
Locations (60):
- United States (60):
  - Horizon Research Group, Inc./Alabama Orthopedic Clinic, Mobile, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Global Research, Anaheim, California
  - Catalina Research Institute, LLC, Chino, California
  - Synergy Clinical Research Center of Escondido, Escondido, California
  - Adam D. Karns MD, Los Angeles, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Clinical Research of West Florida - Clearwater, Clearwater, Florida
  - Century Clinical Research, Inc., Daytona Beach, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Florida Health Center, Fort Lauderdale, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Drug Study Institute, Jupiter, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - NEMA Research, Inc., Naples, Florida
  - Compass Research, LLC, Orlando, Florida
  - Peninsula Research, Ormond Beach, Florida
  - Gold Coast Research, L.L.C., Plantation, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clinical Research of West Florida - Tampa, Tampa, Florida
  - National Pain Research Institute, LLC, Winter Park, Florida
  - Atlanta Research Center, Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Taylor Research, LLC, Marietta, Georgia
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - International Clinical Research Institute, Inc., Overland Park, Kansas
  - Willis-Kinghton Physician Network/River Interventional Pain Specialist, Bossier City, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Best Clinical Trials, Inc., New Orleans, Louisiana
  - River Cities Clinical Research Center, Shreveport, Louisiana
  - MedVadis Research Corp., Watertown, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Office of Robert Kaplan, DO, Las Vegas, Nevada
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - PharmQuest, LLC, Greensboro, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Plains Medical Clinic, LLC, Fargo, North Dakota
  - Clinical Inquest Center, Ltd., Beavercreek, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Optimed Research, Ltd., Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - NPC Research, Oklahoma City, Oklahoma
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - FutureSearch Clinical Trials - Austin, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Advanced Clinical Research of Houston, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - Clinical Investigations Specialists, Inc., Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1633 subjects screened, a total of 752 subjects were enrolled into the open-label (OL) titration phase. Subjects who completed the OL titration phase (462) were eligible for randomization in the double-blind (DB) treatment phase.
Groups:
- OL Buprenorphine HCl Buccal Film: Buprenorphine hydrochloride (HCl) buccal film, 75, 150, 300, or 450 µg, applied to the buccal mucosa every 12 hours for up to 8 weeks in the open-label titration phase
- DB Buprenorphine HCl Buccal Film: Buprenorphine HCl buccal film, 150, 300, or 450 µg, applied to the buccal mucosa every 12 hours for 12 weeks in the double-blind treatment phase
- DB Placebo Film: Placebo buccal film applied to the buccal mucosa every 12 hours for 12 weeks in the double-blind treatment phase
Period: Open-label Titration Phase
Arm/Group | OL Buprenorphine HCl Buccal Film | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Started | 752 | 0 | 0
Completed | 462 | 0 | 0
Not Completed | 290 | 0 | 0
Not completed — Adverse Event | 109 | 0 | 0
Not completed — Lack of Efficacy | 33 | 0 | 0
Not completed — Withdrawal by Subject | 34 | 0 | 0
Not completed — Protocol Violation | 24 | 0 | 0
Not completed — Lost to Follow-up | 22 | 0 | 0
Not completed — Other | 68 | 0 | 0
Period: Double-blind Treatment Phase
Arm/Group | OL Buprenorphine HCl Buccal Film | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Started | 0 (All subjects completing OL titration in the previous period were randomized to a DB treatment.) | 230 (Subjects were randomized to DB treatment after completing OL titration in the previous period.) | 232 (Subjects were randomized to DB treatment after completing OL titration in the previous period.)
Completed | 0 | 176 | 174
Not Completed | 0 | 54 | 58
Not completed — Adverse Event | 0 | 13 | 7
Not completed — Lack of Efficacy | 0 | 8 | 23
Not completed — Withdrawal by Subject | 0 | 11 | 8
Not completed — Protocol Violation | 0 | 7 | 10
Not completed — Lost to Follow-up | 0 | 4 | 9
Not completed — Withdrawal due to opioid withdrawal | 0 | 3 | 1
Not completed — Not exposed to DB study medication | 0 | 1 | 0
Not completed — Other | 0 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Analysis based on intent-to-treat (ITT) population; all randomized subjects who received at least 1 dose of double-blind study medication. One (1) subject did not receive double-blind study medication and an additional 41 subjects from 1 site were excluded from the population.
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film | Total
Number analyzed (Participants) | 209 | 211 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 186 | 366
  >=65 years | 29 | 25 | 54
Age, Continuous [Median (Full Range); unit: years] | 52.0 [22 to 82] | 49.0 [19 to 78] | 51.0 [19 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 107 | 124 | 231
  Male | 102 | 87 | 189
Region of Enrollment [Number; unit: participants]
  United States | 209 | 211 | 420

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Average Daily Pain Intensity Scores
Description: Change in pain intensity = average of daily pain scores from the last 7 days prior to Week 12 visit - average of daily pain scores for the last 7 days prior to randomization. Average pain intensity over the last 24 hours was rated on an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Baseline, Week 12
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication. One (1) subject did not receive double-blind study medication and an additional 41 subjects from 1 site were excluded from the population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 209 | 211
units on a scale | 0.94 (1.846) | 1.59 (2.040)
Statistical Analysis 1: Comparison: DB Buprenorphine HCl Buccal Film vs DB Placebo Film; Test type: Superiority or Other; p = 0.0012, ANCOVA; Median Difference (Net) = -0.67, 95% CI 2-sided [-1.07 to -0.26]

2. Secondary Outcome: Number of Participants With Response to Treatment (Responder) Using NRS Scale
Description: Responders are subjects who achieve a relative reduction in pain intensity from the start of open-label titration to Week 12 in double-blind treatment. Average pain intensity over the last 24 hours was rated on an 11-point NRS ranging from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Prior to open-label titration to Week 12 in double-blind treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 209 | 211
participants
  Responders with ≥30% pain reduction | 131 | 99
  Responders with ≥50% pain reduction | 86 | 69
Statistical Analysis 1: Comparison: DB Buprenorphine HCl Buccal Film vs DB Placebo Film; Responders with ≥30% pain reduction; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel; Stratified by stratum (dose level)
Statistical Analysis 2: Comparison: DB Buprenorphine HCl Buccal Film vs DB Placebo Film; Responders with ≥50% pain reduction; Test type: Superiority or Other; p = 0.0754, Cochran-Mantel-Haenszel; Stratified by stratum (dose level)

3. Secondary Outcome: Number of Subjects With Rescue Medication Use
Description: Use of analgesic rescue medication recorded in subject diary.
Time Frame: Week 1 to Week 12 in double-blind treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 209 | 211
participants
  Week 1 | 123 | 140
  Week 2 | 112 | 132
  Week 3 | 85 | 107
  Week 4 | 81 | 98
  Week 5 | 76 | 92
  Week 6 | 74 | 94
  Week 7 | 73 | 85
  Week 8 | 64 | 85
  Week 9 | 67 | 82
  Week 10 | 60 | 81
  Week 11 | 62 | 72
  Week 12 | 56 | 72

4. Secondary Outcome: Time to Optimal Dose of Open-label Study Medication
Description: Overall time to reach the "optimal" dose of study medication required to progress to double-blind treatment.
Time Frame: Up to 8 weeks in open-label titration
Population: Analysis based on randomized subjects in the Safety population; all subjects who received at least 1 dose of study medication and were randomized into double-blind treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OL Buprenorphine HCl Buccal Film
Number analyzed (Participants) | 462
days | 17.1 (7.77)

5. Secondary Outcome: Percentage of Participants With Treatment Failure in the Double-blind Treatment Phase (up to 12 Weeks)
Description: Treatment failure is defined as study discontinuation due to lack of efficacy or discontinuation due to adverse events in the double-blind treatment phase.
Time Frame: Baseline to treatment failure or end of double-blind treatment phase (up to 12 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 209 | 211
percentage of participants | 9.6 | 14.2

6. Secondary Outcome: Patient Global Impression of Change
Description: Subjects assessed their change in activity limitations as they relate to their painful condition since beginning treatment using the Patient Global Impression of Change (PGIC) questionnaire, a 7-point scale ranging from 1 (no change [or condition has got worse]) to 7 (a great deal better, and a considerable improvement that made all the difference)
Time Frame: Week 12
Population: Analysis based on Patient-Reported Outcomes (PRO) population; randomized subjects who received at least 1 dose of double-blind medication and had at least 1 post-dose assessment on PRO measures. Subjects from 1 site excluded from population (41). Includes only participants with PGIC assessment at week 12 (n=198 buprenorphine and n=194 placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 198 | 194
units on a scale | 4.5 (1.75) | 3.9 (1.99)

7. Secondary Outcome: Change From Baseline to Week 12 in Roland Morris Disability Questionnaire
Description: Subjects assess disability due to back pain using the Roland Morris Disability Questionnaire (RMDQ) consisting of 24 statements of disability. The score of the RMDQ is the total number of items checked, ranging from 0 to 24 with higher scores indicating greater disability.
Time Frame: Baseline, Week 12
Population: Analysis based on PRO population; randomized subjects who received at least 1 dose of double-blind study medication and had at least 1 post-dose assessment on PRO measures. Subjects from 1 site are excluded from the population (41). Includes only participants with RMDQ assessment at week 12 (n=193 buprenorphine and n=189 placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 193 | 189
units on a scale | 0.6 (5.37) | 1.2 (5.75)

8. Secondary Outcome: Change From Baseline to Week 12 in Medical Outcomes Score Sleep Subscale
Description: Medical Outcomes Score (MOS) Sleep Scale uses 12 items to measure 6 dimensions of sleep (sleep disturbance, somnolence, sleep adequacy, snoring, awaken short of breath or headache, and quantity of sleep/optimal sleep) and an overall sleep problems index score. The scores of the dimensions (except quantity of sleep/optimal sleep) and of the sleep problem index range on a 0 to 100 scale, with higher scores reflecting more of the attribute implied by the name (eg, greater sleep disturbance, greater adequacy of sleep).
Time Frame: Baseline, Week 12
Population: Analysis based on PRO population; randomized subjects who received at least 1 dose of double-blind study medication and had at least 1 post-dose assessment on PRO measures. Subjects from 1 site are excluded from the population (41). Includes only participants with MOS assessment at week 12 (n=199 buprenorphine and n=194 placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 199 | 194
units on a scale
  Sleep problems index | -0.23 (8.274) | 0.10 (8.480)
  Sleep disturbance | -1.43 (12.405) | -1.68 (12.515)
  Somnolence | 0.90 (15.823) | 0.14 (17.381)
  Sleep adequacy | 1.71 (19.204) | 6.19 (19.285)

ADVERSE EVENTS:
Time Frame: From informed consent at screening through 14 days after last dose in the double-blind treatment phase (up to 24 weeks)
Description: Analysis based on Safety population; all enrolled subjects who received at least 1 dose of study drug in the respective period (open-label titration and double-blind treatment)
Groups:
- OL Buprenorphine HCl Buccal Film: Buprenorphine HCl buccal film, 75, 150, 300, or 450 μg, applied to the buccal mucosa every 12 hours for up to 8 weeks in the open-label titration treatment phase
- DB Buprenorphine HCl Buccal Film: Buprenorphine HCl buccal film, 150, 300, or 450 μg, applied to the buccal mucosa every 12 hours for 12 weeks in the double-blind treatment phase
- DB Placebo Film: Placebo buccal film, applied to the buccal mucosa every 12 hours for 12 weeks in the double-blind treatment phase
Arm/Group | OL Buprenorphine HCl Buccal Film | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Serious Adverse Events (participants affected / at risk) | 4/749 | 3/229 | 1/232
Other Adverse Events (participants affected / at risk) | 443/749 | 43/229 | 31/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL Buprenorphine HCl Buccal Film (N=749) | DB Buprenorphine HCl Buccal Film (N=229) | DB Placebo Film (N=232)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL Buprenorphine HCl Buccal Film (N=749) | DB Buprenorphine HCl Buccal Film (N=229) | DB Placebo Film (N=232)
Constipation (Gastrointestinal disorders) | 97 (105) | 9 (9) | 6 (6)
Nausea (Gastrointestinal disorders) | 373 (669) | 23 (32) | 17 (23)
Vomiting (Gastrointestinal disorders) | 58 (62) | 9 (10) | 1 (1)
Dizziness (Nervous system disorders) | 48 (52) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 60 (62) | 5 (5) | 8 (9)
Somnolence (Nervous system disorders) | 52 (56) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI and Institution reserve the right to publish and present the results of the work performed provided that Institution and/or PI submits a copy of any proposed publication to Sponsor's agent for review and comment at least 90 days in advance of its presentation or submission for publication. In addition, if Sponsor's agent requests, Institution and/or PI will withhold publication or presentation for an additional 60 days to allow for establishing and preserving its proprietary rights.